CLINICAL TRIAL: NCT02002364
Title: A Comparison Between Flexible Single Use Endoscopes (Ambu aScopes) and Reusable Flexible Endoscopes Used as a Standard of Car When Intubation the Trachea Via an Aura-I Supraglottic Airway Device
Brief Title: Comparison of a Single Use (Ambu aScope) and a Reusable Flexible Optical Scope for Intubation Through a Supraglottic Airway Device (Aura-i)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Consultant anaesthetist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Journal nr. H-3-2012-001
Record Dates: First submitted 2013-11-24; First posted 2013-12-05 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: General Anesthesia
Keywords: tracheal intubation
MeSH Terms: interventions — Intubation, Intratracheal

ARMS (2):
- Single use flexible optical scope (Active Comparator): Single use flexible optical scope , Ambu aScope
  Interventions: Procedure: tracheal intubation
- Multiple use flexible optical scope (Active Comparator): Multiple use flexible optical scope
  Interventions: Procedure: tracheal intubation

INTERVENTIONS:
Procedure: tracheal intubation

SUMMARY:
In patient who are predicted to be difficult to intubate with a standard direct laryngoscope well use flexible optical intubation via a supraglottic airway devise (the Ambu Aura-i). Patients are randomly assigner to a single- or a multiple- use flexible optical scope.

We hypothesize that intubation is obtained equally effective with both types of flexible scopes

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3 and evaluated pre-operatively and found suitable for tracheal intubation with a flexible optical scope via the SAD and scheduled for elective surgery/anesthesia and are conscious about their rights and consequences of participating in the study.
* The patient must have one or two of the following predictors of difficult tracheal intubation:

  1. Modified Mallampati score > 2 (= "no parts of the Uvula is visible")
  2. a thyromental distance of less then or equal to 6.5 cms
  3. Combined movement in head and neck < 90 degrees
  4. Mouth-opening less the 4 cm (but must be larger then 2.5 cm)
  5. Inability to protrude the teeth n the lower jaw beyond the upper incisors
  6. BMI > 40 combined with a neck-circumference > 43 cms
  7. Upper-lip-bite-test > 2
  8. Previous difficult intubation or laryngoscopy (If more then two criteria are fulfilled the patient should be considered intubated awake instead. . But the upper-lip-bite-test and the prognation-beyond the incisors test represents a similar thing, namely the inability to sub-luxate the lower jaw, the if both these findings are positive it is only considered as counting for one.

Exclusion Criteria:

* ASA physical status 4 or 5
* contraindications for use of the SAD
* Patients in whom intubation via a SAD has previously failed
* Patients at risk of aspiration from the gastrointestinal channel
* diseases in mouth, pharynx or larynx that precludes the use of a SAD
* Patients in whom the cricothyroid membrane cannot be localized preanaesthetically
* Patients in whom the doctor making the pre-anaesthetic evaluation finds in need of an awake intubation
* Patients with possible Creutzfeldt-Jacobs disease or contraindication against the use of non-autoclavable equipment r risk of cross contamination with prions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Duration of intubation. From the endoscope enters the supraglottic-airway-device to CO2-curve is seen | Measured during tracheal intubation at induction of anesthesia

SECONDARY OUTCOMES:
Number of attempts at placing the supraglottic-airway-device (SAD) | From anesthesia induction and the following 10 minutes during securing of the airway
  an attempt is defined as the tip of the SAD passing the upper front teeth
number of attempts at placing the flexible endoscope in the trachea | From anesthesia induction and the following 10 minutes
number of attempts at intubation | From anesthesia induction and during the following 10 minutes during airway management
  An intubation attempt starts when the tip of the endotracheal tube passes the entrance to the SAD
Total time for placement of SAD and endoscopy and intubation | During induction of anesthesia and the following 10 minutes during airway management
The best glottic view obtained | After anesthesia induction and during the following 10 minutes during airway management
The ease of passage of the flexible endoscope via the SAD | During induction and airway management
The anesthesiologists' satisfaction with the procedure | During induction of anesthesia and within the 30 minutes hereafter
The quality of the endoscopically obtained image | During induction of anesthesia and the following 10 minutes during airway management
Postoperative sore throat, dysphonia or dysphagia one hour after extubation | AT the time 1 hour after extubation of the trachea

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Rigshospitalet, Denmark, Copenhagen, Denmark
- Service d'anesthesie-reanimation 1 avenue Moliere Hopiatl de Hautepierre, Strasbourg, France